CLINICAL TRIAL: NCT04072172
Title: Microcautery Evaluation for Treatment of Leg Spiders
Brief Title: Microcautery for the Treatment of Spider Leg Veins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa M. Selim, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Micro-cautery for leg veins
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Microcautery for Leg Veins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female with leg spider veins (Experimental): Females at the age of 20 to 45 not known diabetics or hypertensive complaining of leg spider veins.
  Interventions: Device: Mole Freckle Pen

INTERVENTIONS:
Device: Mole Freckle Pen — Insulated micro steel needle use current: 5V / 1A of 5-speed free adjustment.5

SUMMARY:
To Evaluate the role of micro-cauterization use in the treatment and disappearance of spider leg veins.

DETAILED DESCRIPTION:
Spider veins on the lower limbs are very common and have been reported to be presented in 41% of women over 50 years old. Sclerotherapy as a traditional treatment for spider veins has a low cost, though it may have adverse sequelae. Lasers have shown fewer but still substantial complications as well.1 Spider veins are small superficial veins that widen and become visible, often on the legs and most cutaneous spider veins are abnormalities of the horizontal vascular skin plexus or capillary loops.2 Spider leg veins are composed of a feeder vessel and ectatic venous sprouts in the reticular dermis. Their depth is between 180 µm and 1 mm in the skin.3 Spider veins may have a diameter that reaches several millimetres and can be blue, purple or red and may appear in the form of thin lines, webs or branches.4 There is a scarce available data from literature about the role of micro-cauterization in the treatment of spider veins. The micro-cauterization is an alternative in management of spider veins that delivered via Mole Freckle Pen German Technology.4 Cautery is a safe and effective tool for the treatment of superficial and small skin lesions. It is simple, cheap, and requires minimal training and the results are usually satisfactory Technology Specifications with insulated micro steel needle use current: 5V / 1A of 5-speed free adjustment.5 The current study aims to evaluate the role for micro-cauterization in the treatment and disappearance of spider leg veins.

ELIGIBILITY:
Inclusion Criteria:

* were patients with spider veins of less than 2.0 mm in diameter.

Exclusion Criteria:

* were patients with diabetes, anticoagulation therapy and/or patients with a known history of keloids

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Short term results after 3 weeks. | 3 weeks
  Compare between the shape of spider leg veins pre and post the cauterization session depending on standard Oriented photos taken pre and post.

SECONDARY OUTCOMES:
Long term results after 3 months. | 3 months
  Study, monitor and evaluate the long term results of the cautery session after 3 months and if there is any reappearance of the spider veins with a standard Oriented photos taken.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa M. Selim, Resident, Principal Investigator — Assiut University